CLINICAL TRIAL: NCT04884386
Title: Effects of WALKBOT-G Robot-assisted Gait Training on Anticipatory Posture Adjustment Function and Balance With Bilateral Spastic and Hemiplegic Cerebral Palsy: A Single-blind Randomized Controlled Trial
Brief Title: Effects of WALKBOT-G Robot-assisted Gait Training on Anticipatory Posture Adjustment Function and Balance With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Hyun-Joong Kim, collaborator, Sahmyook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2-1040781-A-N-012021048HR
Record Dates: First submitted 2021-05-08; First posted 2021-05-13 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Cerebral Palsy; Spastic Hemiplegic Cerebral Palsy; Bilateral Spastic Cerebral Palsy; Gait Disorders, Neurologic
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robot-assisted gait training (Experimental)
  Interventions: Device: robot-assisted gait training; Behavioral: conventional locomotion therapy
- conventional locomotion therapy (Active Comparator)
  Interventions: Behavioral: conventional locomotion therapy

INTERVENTIONS:
Device: robot-assisted gait training — RAGT, WALKBOT-G, is a walking training equipment that can reproduce natural motions by adjusting the leg length and adjusting the motion with the actuator of the ankle joint.
  Arms: robot-assisted gait training
Behavioral: conventional locomotion therapy — locomotion exercise, postural control training, balance training, electrotherapy

SUMMARY:
In children with cerebral palsy, the quality of walking decreases due to a decrease in the ability to control limbs, including walking, and coordination among various activities of daily living due to a decrease in functional independence and quality of life. Gait disorder is one of the important therapeutic goals of children with cerebral palsy, and recently robot-assisted gait training (RAGT) induces changes in brain plasticity, so it will help improve gross motor control and coordination control.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 6-12 years or younger who have not received botulinum toxin or surgery within 3 months before the study
* Patients diagnosed with Bilateral Spastic Cerebral Palsy
* Patients diagnosed with Spastic Hemiplegic Cerebral Palsy

Exclusion Criteria:

* Children who cannot understand and follow orders
* Children with stiffness in the lower limbs corresponding to the Modified Ashworth Scale (MAS)> 3
* Patients who wear a robot and walk without affecting contractures, deformities, or skin problems
* Infants with cardiovascular instability and mild scoliosis with a cobb's angle of 30 degrees or more

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2021-06-12 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
muscle activation | Change from baseline muscle activation at 4 weeks
  Measure muscle activity of Sternocleidomastoid, C4 Cervical Paraspinals, L5 Paraspinals, Rectus Femoris, Medial Hamstring, and Soleus during functional reach test. Surface electromyograph(EMG)(Mini Wave Infinity Waterproof, Cometa Systems, Italy, 2017) was used to measure muscle activity, and analysis software(Myoresearch XP Master 1.07, Noraxon, USA, 2011) was used for EMG analysis. The sampling rate was set to 2000 Hz. The EMG raw data was quantified as 150 ms after applying full wave rectification, and filtering was performed in the range of 20 to 450 Hz using a digital band-pass filter (Lancosh FIR). do

CONTACTS AND LOCATIONS:
Locations (1):
- Ez rehabilitation medical center, Yongin-si, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
I plan to decide after the study is over.